CLINICAL TRIAL: NCT03141203
Title: Phase I/II Study to Determine the Maximum Tolerated Dose and Activity of the Combination of Romidepsin and Carfilzomib in Relapsed or Refractory Peripheral T-cell Lymphoma
Brief Title: Evaluation of the Combination of Romidepsin and Carfilzomib in Relapsed/Refractory Peripheral T Cell Lymphoma Patients
Acronym: RomiCar
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Bloodwise (Other); Celgene (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_13-107; 2013-001879-20 (EudraCT Number)
Record Dates: First submitted 2017-02-21; First posted 2017-05-05 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — romidepsin; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Dose Level 1 (Experimental): 8mg/m2 Romidepsin (administered on days 1, 8, 15) and 20/36mg/m2 Carfilzomib (administered days 1, 2, 8, 9, 15, 16) over 8 cycles of treatment.
  Carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.
  Interventions: Drug: Romidepsin; Drug: Carfilzomib
- Dose Level 2 (starting dose) (Experimental): 10mg/m2 Romidepsin (administered on days 1, 8, 15) and 20/36mg/m2 Carfilzomib (administered days 1, 2, 8, 9, 15, 16) over 8 cycles of treatment.
  Carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.
  Interventions: Drug: Romidepsin; Drug: Carfilzomib
- Dose Level 3 (Experimental): 10mg/m2 Romidepsin (administered on days 1, 8, 15) and 20/45mg/m2 Carfilzomib (administered days 1, 2, 8, 9, 15, 16) over 8 cycles of treatment.
  Carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.
  Interventions: Drug: Romidepsin; Drug: Carfilzomib
- Dose Level 4 (Experimental): 12mg/m2 Romidepsin (administered on days 1, 8, 15) and 20/45mg/m2 Carfilzomib (administered days 1, 2, 8, 9, 15, 16) over 8 cycles of treatment.
  Carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.
  Interventions: Drug: Romidepsin; Drug: Carfilzomib
- Dose Level 5 (Experimental): 12mg/m2 Romidepsin (administered on days 1, 8, 15) and 20/56mg/m2 Carfilzomib (administered days 1, 2, 8, 9, 15, 16) over 8 cycles of treatment.
  Carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.
  Interventions: Drug: Romidepsin; Drug: Carfilzomib
- Dose Level 6 (Experimental): 14mg/m2 Romidepsin (administered on days 1, 8, 15) and 20/56mg/m2 Carfilzomib (administered days 1, 2, 8, 9, 15, 16) over 8 cycles of treatment.
  Carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.
  Interventions: Drug: Romidepsin; Drug: Carfilzomib

INTERVENTIONS:
Drug: Romidepsin — 10mg vial for Injection
  Other Names: Istodax
Drug: Carfilzomib — 60mg vial for injection
  Other Names: Kyprolis

SUMMARY:
This is a multicentre phase I/II trial looking at the combination of romidepsin and carfilzomib.

The aim of the phase I part is to determine the maximum tolerated dose (MTD) of the combination. This part will recruit up to 27 patients, plus possibly an additional 3 patients at the MTD.

The aim of the phase II part is to assess the activity of the combination at the maximum tolerated dose in 28 patients (including at least 6 patients treated at the MTD from phase I).

Patients will receive 8 cycles of romidepsin with carfilzomib and response will be assessed every second cycle. Patients will be followed up for progression and survival until the end of the trial.

DETAILED DESCRIPTION:
This is a prospective, single arm, phase I/II, multicentre, dose finding study of romidepsin in combination with carfilzomib.

The aim of the phase I is to establish the MTD of the combination using a restricted two-stage CRM. The MTD is defined as the dose level that is closest to the level at which 25% of patients experience a DLT over the first cycle of treatment.

The intention in phase I is to evaluate the DLT-inducing effects of doses in cohorts of patients. Patients will be treated in cohorts at a dose level and each patient will be evaluated for presence or absence of DLT. In stage I, the first cohort of 3 patients will be enrolled at the starting dose, i.e. dose level 2. If none experiences a DLT, the next cohort of 3 patients will be recruited at the next higher level, i.e. dose level 3. This escalation routine will continue until the first DLT is observed or the maximum recruitment for stage I is reached. As soon as the first DLT is observed, dose escalation and de-escalation will be guided by the CRM design that will recommend the dose believed to have associated DLT-rate closest to 25%. If the trial escalates, each dose below the newly tested dose is regarded as being tolerable.

In stage II, we will consider variable cohort sizes of up to eight patients. Patients are screened for eligibility before they are formally registered. During screening, we expect it to transpire that some patients will be ineligible. To maximise recruitment and reduce trial suspension period between cohorts in this rare disease, we will allow for the flexibility of variable cohort sizes by screening cohorts of up to eight patients. We will allocate screening slots so that the sum of: a) the number of patients already receiving treatment in the current cohort; and (b) the number of patients in screening; does not exceed eight. If a patient is screened and proves to be eligible, they will be recruited to the trial. The first three patients in a cohort will receive the dose-level allocated to the cohort. Patients who are inevaluable, as described immediately above, can be replaced. If the fourth to eighth patients are recruited to a cohort and the dose allocated to the cohort is not yet regarded as tolerable, the fourth to eighth patients will receive the next dose-level below. Otherwise, they will receive the same dose level as the previous patients in the cohort. The aim of the described strategy is to maximise recruitment but not expose more than three patients to a dose that has not yet been demonstrated tolerable. The model will be updated regularly and subsequent recommended doses will be assigned to patients iteratively until the maximum sample size is reached, or the trial is stopped early because there is a high chance that the lowest dose is too toxic. It is expected that the CRM will likely allocate patients to the eventual MTD at the later stage of the trial as more data accumulate. Recruitment will be permitted to continue seamlessly to the Phase II component at the latest recommended MTD dose, in consultation with the Trial Safety Committee, unless it is considered necessary to halt recruitment The initial guess of MTD is at dose combination level 4, however to exercise caution, dose level 2 is defined as the starting dose level.

Dose Levels

1. 8mg/m2 Romidepsin (days 1, 8, 15), 20/36mg/m2 Carfilzomib (days 1, 2, 8, 9, 15, 16)
2. (Starting dose) 10mg/m2 Romidepsin (days 1, 8, 15), 20/36mg/m2 Carfilzomib (days 1, 2, 8, 9, 15, 16)
3. 10mg/m2 Romidepsin (days 1, 8, 15), 20/45mg/m2 Carfilzomib (days 1, 2, 8, 9, 15, 16)
4. 12mg/m2 Romidepsin (days 1, 8, 15), 20/45mg/m2 Carfilzomib (days 1, 2, 8, 9, 15, 16)
5. 12mg/m2 Romidepsin (days 1, 8, 15), 20/56mg/m2 Carfilzomib (days 1, 2, 8, 9, 15, 16)
6. 14mg/m2 Romidepsin (days 1, 8, 15), 20/56mg/m2 Carfilzomib (days 1, 2, 8, 9, 15, 16) For all dose levels, the carfilzomib dose will be 20mg/m2 for the first 2 doses (i.e. day 1 and 2 of cycle 1), rising to the target dose for subsequent doses and cycles.

Once the MTD is defined, patients recruited at a lower dose may receive the MTD for any subsequent cycles of treatment at the discretion of the treating Investigator and the Chief Investigator.

The phase II component will aim to provide a preliminary estimate of activity in 28 patients at the MTD combination established in phase I. The phase II component is based on A'Hern's single arm, single stage design and would utilise patients allocated to the MTD in phase I. Patients will be recruited over a 36-month period and will receive a minimum of 8 cycles of treatment. Patients will continue to be followed up for progression and survival until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years of age
* Life expectancy > 12 weeks
* ECOG performance status ≤ 2
* Relapsed or refractory peripheral T-cell lymphoma including the following histologies: peripheral T-cell lymphoma not otherwise specified, angioimmunoblastic T-cell lymphoma, anaplastic large cell lymphoma, enteropathy associated T-cell lymphoma, extranodal NK/T-cell lymphoma, transformed mycosis fungoides, hepatosplenic T-cell lymphoma [For all relapsed patients, relapse must be confirmed by tissue biopsy (or bone marrow trephine if no other tissue available). For refractory patients, a biopsy must have been obtained within the last 6 months and preferably to confirm refractory disease. In rare cases (such as when re-biopsy is not possible), the initial diagnostic biopsy may be accepted, provided that the patient has been reviewed at the local MDT who agreed that the presentation is consistent with relapsed/refractory T cell lymphoma, and this has been documented.]
* Failed at least 1 prior therapy (but no upper limit of prior regimens)
* Patients MAY have had a prior allogeneic stem cell transplant but must not require systemic immunosuppression for graft-versus-host disease (local treatments are permitted)
* Adequate haematopoietic reserve (Hb ≥ 9g/dl, neutrophils ≥ 1.0x10^9/l and platelets ≥ 100x10^9/l or ≥ 75x10^9/l if marrow involvement documented)
* Adequate liver function (bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless due to Gilbert's syndrome), AST / ALT ≤ 2x ULN)
* Adequate renal function (creatinine clearance ≥ 20ml/min as assessed by Cockcroft and Gault calculation)
* Serum potassium ≥ 3.8 mmol/l, calcium ≥ 2.2 mmol/l and magnesium ≥ LLN prior to trial entry (supplements permitted)
* CT measurable disease with at least 1 lesion having short axis > 1.5cm or splenomegaly > 14cm in cranio-caudal length attributable to relapsed lymphoma
* Ability to give informed consent

Exclusion Criteria:

* Persistent treatment related toxicities of CTCAE v4.0 grade ≥ 2
* Previous treatment with histone deactylase inhibitor or proteasome inhibitor
* Need for any other concurrent anti-cancer drug (apart from corticosteroids at a dose equivalent to prednisolone ≤ 7.5mg daily). A steroid prephase may be used but should be stopped by the first day of cycle 1.
* Concurrent medical illness deemed by the investigator as uncontrolled and/or clinically significant
* Previous systemic malignancy within the last 3 years unless treated with curative intent with no sign of recurrence. Other exceptions include non-melanotic skin cancer or carcinoma in-situ of the uterine cervix
* Co-existing active infection requiring parenteral antibiotics
* Patients unable to swallow oral medication
* Active infection with HIV, hepatitis B or hepatitis C
* Radiotherapy* (except for palliative reasons), endocrine therapy, immunotherapy or use of other investigational agents within 28 days prior to trial entry (or a longer period depending on the defined characteristics of the agents used, please contact the trials office for confirmation). *Limited field radiotherapy to an isolated lesion in bone or soft tissue must be completed 2 weeks prior to trial entry
* Major surgery within 4 weeks of trial entry
* Patients with proven CNS involvement
* QTc interval of >450ms or patients taking medications that significantly prolong the QT interval
* Patients taking any inhibitors or strong inducers of CYP3A4, with the exception of dexamethasone.
* Clinically significant cardiac disease ≥ NYHA Class III, symptomatic ischaemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction within 6 months of trial entry
* Pregnant and lactating patients (patients of childbearing potential must have a negative pregnancy test prior to study entry and within 7 days prior to the start of treatment. Postmenopausal females (> 45 years old and without menstruation for > 1 year) and surgically sterilised females are exempt from a pregnancy test)
* Patients and partners of childbearing potential not willing to use effective contraception during and for 3 months after therapy
* Concurrent Pulmonary Hypertension
* Left Ventricular Ejection Fraction (LVEF) of <40%

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of the combination of romidepsin and carfilzomib | Cycle 1 (each cycle is 28 days)
  MTD as determined by the continual reassessment model (CRM) with a predefined target Dose Limiting Toxicity (DLT) probability of 25%
Best overall response rate (PR + CR) at the MTD | Data will be collected over the first 8 cycles of therapy (each cycle is 28 days)
  Assessed using the International response criteria

SECONDARY OUTCOMES:
Toxicity of the combination of romidepsin and carfilzomib | Adverse events information will be collected throughout the 36 month recruitment period of the trial and during the one year follow up period
  Assessed using CTCAE v4
Best overall response at the MTD | Information relating to this outcome will be collected up to and including the one year follow-up time point
  Assessed using International response criteria
Maximum percentage change in the radiological sum of the product of the diameters from baseline, assessed using the Revised Response Criteria for Malignant Lymphoma | Information relating to this outcome will be collected up to and including the one year follow-up time point
  Assessed on suitable target and non-target lesions
Duration of response from time of first documented response until relapse or progression | Information relating to this outcome will be collected up to and including the one year follow-up time point
Progression free survival | Information relating to this outcome will be collected up to and including the one year follow-up time point
Overall survival | Information relating to this outcome will be collected up to and including the one year follow-up time point

CONTACTS AND LOCATIONS:
Overall Officials: Graham Collins, MBBS DPhil, Principal Investigator — Churchill Hospital, Oxford, UK
Locations (13):
- United Kingdom (13):
  - Queen Elizabeth Hospital, Birmingham
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - Guy's Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hospitals, London
  - Christie Hospital, Manchester
  - Nottingham University Hospitals, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No